CLINICAL TRIAL: NCT06011031
Title: Mechanical and Biological Assessment of Two Different Attachment Materials in Maxillary Implant Retained Overdenture In-Vivo Study
Brief Title: Assessment of Novaloc and Locator Attachment Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU- Rec ID 032117
Record Dates: First submitted 2023-07-21; First posted 2023-08-25 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-07

CONDITIONS: Completely Edentulous Maxilla
Keywords: implant overdenture; maxilla; novaloc; locator; peek

STUDY DESIGN:
Intervention Model Description: This is a Randomized Clinical Trial (phase IV) as it will compare two types of attachment systems (a new one with an old one), assess the effects of both types, and state which one is better.
Who Masked: Investigator
Masking Description: all selected patients were restored with a complete denture prosthesis and then wer devided using random allocation software into 2 groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novaloc attachment (Experimental): a newly developed device "novaloc attachment system"made of peek material and amorphous diamond like carbon.
  Interventions: Device: Novaloc attachment
- locator attachment (Active Comparator): a device with low-profile attachment used in cases of limited inter arch distance, provides excellent retention, possesses a self-aligning property and allow correction of implant divergence up to 20 degrees
  Interventions: Device: Locator attachment

INTERVENTIONS:
Device: Novaloc attachment — Each patient will be restored with 4 implants retained maxillary overdenture with the assigned attachment
  Arms: Novaloc attachment
Device: Locator attachment — Each patient will be restored with 4 implants retained maxillary overdenture with the assigned attachment
  Arms: locator attachment

SUMMARY:
The aim of the current study is to assess the effect of two types of attachments (Locator, Novaloc) on the supporting structures both mechanically using stress strain analysis and biologically through measuring bone height using cbct.

DETAILED DESCRIPTION:
14 Completely edentulous patients will be divided into two groups each group contains seven patients: Group One: Each patient will be restored with 4 implant retained maxillary overdenture using Peek retention inserts attachment system and Bone Level Ti-Zr implants.

Group Two: Each patient will be restored with 4 implant retained maxillary overdenture using Nylon retention insert attachment system and Bone Level Ti implants.

Bone height in millimeters will then be evaluated around each implant using cone beam computed tomography at the time of placement of attachments, 6 months, 1 year

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patient with u shaped dental arch.
* Systemically free.
* Patients completed all extraction at least 6 months before surgery.
* Patients Tempromandibular joint is free from any disease.
* Patient's mouth opening is proper for accessibility during surgery and implant placement.
* Sufficient bone level (length, and width) at implant placement site.
* Presence of enough bone height at implant site close to the maxillary sinus.
* Absence of sinus pneumatization.

Exclusion Criteria:

* Heavy smoker.
* Patients with bone diseases.
* Patients having a history of parafunctional habits.
* Patients with diabetes mellitus.
* Patients on chemotherapy or radiotherapy.
* Patients on any medications that reduce wound healing.
* Patients without sufficient bone level (height, width).
* Patients with sinus pneumatization.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
bone level change around implants | Through study completion an average 1 year.
  measurement of bone height mesial, distal to each implant

SECONDARY OUTCOMES:
patient satisfaction | Through study completion an average 1 year.
  Patient satisfaction was evaluated using a questionnaire based on the visual analog scale (VAS). Patients were asked to mark their answers (amount of satisfaction). The questionnaire was given to the patients in Arabic.Six factors were rated on a 1 to 5 scale (highly satisfied = 5; satisfied = 4; fair = 3; dissatisfied = 2; highly dissatisfied = 1). The sum of the five sub-scores was then calculated, ranging from 5 to 30 (best score = 30, worst score = 5). The low range of scores indicated low satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ibrahim Eid, Prof, Study Director — Ain Shams University; Noha Helmy Nawwar, Prof, Study Director — Ain Shams University; Ahmed Mohamed Osama, Prof, Study Director — Ain Shams University; Fatma Fouad Sadek, AssistantLec, Principal Investigator — Egyptian Russian University
Locations (1):
- Prosthodontics Department Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
once all data is collected, sharing of Study Protocol,Statistical Analysis Plan (SAP),Clinical Study Report (CSR) will be done
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year following publishing
Access Criteria: researchers , students or post graduates